CLINICAL TRIAL: NCT06802016
Title: A Cohort Study of Congenital Bicuspid Aortic Valve
Brief Title: A Study of Chinese Congenital Bicuspid Aortic Valve
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhu zhengbin, deputy chief physician, Ruijin Hospital
Other Study IDs: RJH-BAV
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Bicuspid Aortic Valve (BAV)
Keywords: Bicuspid Aortic Valve; Dilated ascending aorta; Aortic regurgitation; Aortic stenosis; Acoustic cardiography
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Aortic Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood sample at enrollment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pervious studies indicated that the prevalence of bicuspid aortic valve（BAV） might be higher in China. There is a familial predisposition to the development of BAV. The study analyzed epidemiological data on selected BAV and established a BAV cohort to observe disease progression and treatment outcomes.

DETAILED DESCRIPTION:
There is no recognized comprehensive epidemiological data on congenital BAV in China, although findings of BAV is common in clinical practice. In the course of the Venus-A registry clinical study, which was the first Aortic Valve Replacement (TAVR) trial in China, the investigators concluded about 40% of the final enrollment of BAV patients. Since then, an increasing number of scholars have figured out that the prevalence of BAV may be much higher in China than abroad. This study was designed to investigate Gene backgrounds, pathological progress, imaging characteristics of young health BAV participants and their relationships in long-term follow-up. These findings may help to identify high risk individuals with specific gene expression or other features in clinical observation.

ELIGIBILITY:
Inclusion Criteria:

* The patients were aged 14-60 years;
* Definitive diagnosis of BAV by imaging (echocardiography, aortic CTA, cardiac magnetic resonance, etc.)
* Patients were informed about the nature of the study and agreed to participate in all the terms of the study and signed an informed consent form approved by the ethics committee.

Exclusion Criteria:

* Poor patient compliance and inability to complete follow-up visits as required;
* Rheumatic heart valve disease, other organic valve disease.
* Hyperthyroidism, severe anemia, and other factors that significantly affect hemodynamics.
* Other circumstances that the researcher believes should be excluded.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is single-center cohort study. Patients diagnosed with BAV were enrolled in Ruijin Hospital.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
SAVR / TAVR | 5 year
  Indications for surgical or transcatheter aortic valve replacement

SECONDARY OUTCOMES:
Major adverse cardiovascular events(MACE) | 5 year
  Ascending aortic aneurysm or aortic dissection, all-cause death, cardiac death, non-fatal stroke, hospitalization for heart failure

OTHER OUTCOMES:
Synchronized analysis of phonocardiogram and electrocardiogram | 6 or 12 month depending on severity of valves
  Synchronized PCG and ECG data using a wearable cardiac monitoring patch
Echocardiography | 6 or 12 month depending on severity of valves
  Valve morphology, Degree of valve stenosis or regurgitation, Degree of widening of the ascending aorta, Left ventricular ejection fraction(LVEF) changes, Degree of left ventricular hypertrophy or enlargement.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengbin Zhu, MD, PhD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided